CLINICAL TRIAL: NCT01780454
Title: Renal Allograft Tolerance Through Mixed Chimerism
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David Sachs M.D., Director, Transplantation Biology Research Center, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013P000822
Record Dates: First submitted 2013-01-29; First posted 2013-01-31 (Estimated); Results first posted 2020-09-23 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-03

CONDITIONS: End Stage Renal Disease
Keywords: End Stage Renal Disease; Renal Transplant; Bone Marrow Transplant; Tolerance; Chimerism; ESRD
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — siplizumab; Rituximab; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combined Bone Marrow and Kidney Transplantation (Experimental): Conditioning regimen consisting of Rituximab, MEDI-507, Total Body Irradiation, Thymic Irradiation followed by simultaneous bone marrow and kidney transplantation
  Interventions: Drug: MEDI-507; Drug: Rituximab; Radiation: Total Body Irradiation; Radiation: Thymic Irradiation

INTERVENTIONS:
Drug: MEDI-507 — T-Cell Depleting Agent
Drug: Rituximab — B-Cell Depleting Agent
Radiation: Total Body Irradiation — Bone Marrow Depletion
Radiation: Thymic Irradiation

SUMMARY:
This study will examine the safety and effectiveness of a combination kidney and bone marrow transplant from a haplo-identical related donor. An investigational medication and other treatments will be given prior to and after the transplant to help protect the transplanted kidney from being attacked by the body's immune system

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female 18-60 years of age
* Candidate for a living-donor renal allograft with a one haplotype identical donor identified.
* First or second transplant with either a living donor or cadaveric transplant as the first transplant.
* Positive serologic testing for EBV indicating past exposure.

Key Exclusion Criteria:

* ABO blood group-incompatible renal allograft.
* Evidence of anti-HLA antibody within 60 days prior to transplant as assessed by routine methodology (AHG and/or ELISA)
* Positive testing for: HIV, hepatitis B core antigen, or hepatitis C virus or positivity for hepatitis B surface antigen.
* Cardiac ejection fraction < 40% or clinical evidence of insufficiency.
* History of cancer other than basal cell carcinoma of the skin or carcinoma in situ of the cervix.
* Underlying renal disease etiology with a high risk of disease recurrence in the transplanted kidney (such as focal segmental glomerulosclerosis, type I or II nonproliferative glomerulonephritis).
* Prior dose-limiting radiation therapy.
* Abnormal (>2 times lab normal) values for (a) liver function chemistries (ALT, AST, AP), (b) bilirubin, (c) coagulation studies (PT, PTT).
* The presence of any medical condition that the investigator deems incompatible with participation in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-03; Primary Completion 2018-06 (Actual); Study Completion 2020-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. Benedict Cosimi, M.D., Principal Investigator — Massachusetts General Hospital; David Sachs, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Kawai T, Cosimi AB, Sachs DH. Preclinical and clinical studies on the induction of renal allograft tolerance through transient mixed chimerism. Curr Opin Organ Transplant. 2011 Aug;16(4):366-71. doi: 10.1097/MOT.0b013e3283484b2c. PMID 21666482
- [Background] Sachs DH, Sykes M, Kawai T, Cosimi AB. Immuno-intervention for the induction of transplantation tolerance through mixed chimerism. Semin Immunol. 2011 Jun;23(3):165-73. doi: 10.1016/j.smim.2011.07.001. Epub 2011 Aug 11. PMID 21839648
- [Background] Kawai T, Cosimi AB, Spitzer TR, Tolkoff-Rubin N, Suthanthiran M, Saidman SL, Shaffer J, Preffer FI, Ding R, Sharma V, Fishman JA, Dey B, Ko DS, Hertl M, Goes NB, Wong W, Williams WW Jr, Colvin RB, Sykes M, Sachs DH. HLA-mismatched renal transplantation without maintenance immunosuppression. N Engl J Med. 2008 Jan 24;358(4):353-61. doi: 10.1056/NEJMoa071074. PMID 18216355

RESULTS

PARTICIPANT FLOW:
Groups:
- Combined Bone Marrow and Kidney Transplantation: Conditioning regimen consisting of Rituximab, MEDI-507, Total Body Irradiation, Thymic Irradiation followed by simultaneous bone marrow and kidney transplantation
  MEDI-507: T-Cell Depleting Agent
  Rituximab: B-Cell Depleting Agent
  Total Body Irradiation: Bone Marrow Depletion
  Thymic Irradiation
Period: Overall Study
Arm/Group | Combined Bone Marrow and Kidney Transplantation
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Combined Bone Marrow and Kidney Transplantation
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Successful Withdrawal of Immunosuppressive Therapy
Description: The primary endpoint is induction of transient mixed chimerism and renal allograft tolerance without "engraftment syndrome" or "acute kidney injury"
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Bone Marrow and Kidney Transplantation
Number analyzed (Participants) | 2
Participants | 2

2. Secondary Outcome: Number of Participants With Engraftment Syndrome
Description: Constellation of symptoms known "Engraftment Syndrome"
Time Frame: 5 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Bone Marrow and Kidney Transplantation
Number analyzed (Participants) | 2
Participants | 2

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Combined Bone Marrow and Kidney Transplantation
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined Bone Marrow and Kidney Transplantation (N=2)
Dehydration (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined Bone Marrow and Kidney Transplantation (N=2)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-27): https://cdn.clinicaltrials.gov/large-docs/54/NCT01780454/Prot_SAP_000.pdf